CLINICAL TRIAL: NCT05969106
Title: A Study Comparing Tandem Control-IQ With Real-time Continuous Glucose Monitoring (rtCGM) Used Together With Insulin Pens and Insulin Pumps for 18 Months
Brief Title: Tandem Control-IQ Evaluation Regarding Glucose Metrics, Sleep, and Health Economics
Acronym: STARCARE
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Johan Peter Adolfsson, Principal Investigator, Vastra Gotaland Region
Other Study IDs: VastraGotaland - 2022-00332-01
Record Dates: First submitted 2023-06-30; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- rtCGM + MDI: Real-time CGM Dexcom G6 used in parallel to Multiple Daily Injections (MDI)
  Interventions: Device: Tandem Control-IQ
- rtCGM + CSII: Real-time CGM Dexcom G6 used in parallel to freestanding Continuous Subcutaneous Insulin Infusion (CSII)
  Interventions: Device: Tandem Control-IQ
- Tandem Control-IQ: Realtime CGM Dexcom G6 used as part of the Automated Insulin Delivery (AID) system
  Interventions: Device: Tandem Control-IQ

INTERVENTIONS:
Device: Tandem Control-IQ — AID-system

SUMMARY:
To evaluate Tandem Control-IQ compared with rtCGM and insulin pen respectively rtCGM and insulin pump treatment in children and adolescents regarding glucose control, sleep and health economics for 18 months.

DETAILED DESCRIPTION:
In this obesrvational study, the investigators assessed glycemic outcomes, sleep and health economics associated with AID treatment (Tandem Control-IQ) compared with multiple daily insulin injections with rtCGM (MDI+rtCGM) and a standalone insulin pump with rtCGM (CSII+rtCGM). Participants from two clinical sites in Sweden who continuously used one of the three modalities for at least six months were included in the analysis. Inclusion required all participants to use the Dexcom G6 rtCGM sensor for glucose monitoring, which meant only insulin treatment differentiated the three groups. Comparisons were conducted regarding Hemoglobon A1c (HbA1c) at the start of the study and rtCGM-generated glycemic metrics from 1 month before the study started until 18 months. Sleep quality and quantity were assessed using a questionnaire for the persons with diabetes and the caretakers. Indirect and direct costs in all healthcare systems and additional information on sick leaves were collected from the Swedish Social Insurance Agency. Comparisons were then made between the three treatment alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2-19 years at the start
* Diagnosed with Type 1 diabetes
* Min duration three months
* Willingness to participate in the study

Exclusion Criteria:

* Pregnancy
* Unwillingness to share and upload CGM data
* Reluctance to come to visit and to follow protocol
* History of allergic reaction to Dexcom CGM materials or adhesives in contact with the skin.
* Abnormal skin at the anticipated glucose sensor attachment sites(excessive hair, burn, inflammation, infection, rash, and/or tattoo)

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals diagnosed with Type 1 diabetes at two different pediatric diabetes centres.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Glycemic metrics | Change from baseline to 6, 12 and 18 months
  Time in range (TIR), Time below range (TBR) Level 1 and 2, Time above range (TAR) Level 1 and 2, Time in tighter range (TITR)
Sleep | At study completion at 12 months.
  Quantity and quality are defined in the questionnaire. Assessment by a 10-point Likert scale (1= "Worst possible", 10= "Best possible")
Costs - direct | From baseline until study completion at 18 months
  Cost for the insulin administration devices and continuous glucose monitoring devices per person/year (direct). All costa are calculated in Swedish currency (SEK).
Costs - indirect | From baseline until study completion at 18 months
  Cost for comorbidities and all health-care related costs (indirect), including societal costs based on days with sick-leaves (indirect). All costs are calculated in Swedish currency (SEK).
Quality Adjusted Life Year (QALY) | From baseline until study completion at 18 months.
  Quality Adjusted Life Year is estimated for each health state by literature search and for each of the three treatment alternatives. QALY is a generic measure of disease burden, including both the quality and the quantity of life lived. It is used in economic evaluation to assess the value of medical interventions. One QALY equates to one year in perfect health. QALY scores range from 1 (perfect health) to 0 (dead). Thus, a higher value means a better outcome.
Cost/QALY | From baseline until study completion at 18 months.
  Cost/QALY is estimated for each health state by literature search and for each of the three treatment alternatives. Cost/QALY is illustrating the cost per disease burden, including both the quality and the quantity of life lived. It is used in economic evaluation to assess the cost per value of medical interventions. A lower value means a better outcome.
Incremental Cost Efficiency Rate (ICER) | From baseline until study completion at 18 months.
  Based on glucose control cost-effect pairs is generated for Tandem Control-IQ vs. MDI respectively Tandem-Control-IQ vs. CSII. An ICER is calculated by dividing the difference in total costs (incremental cost) by the difference in the chosen measure of health outcome or effect (incremental effect) to provide a ratio of 'extra cost per extra unit of health effect' - for therapy A vs therapy B. A higher value means a better outcome. A prediction is added 10-, 20-, and 30-years ahead. ICER is estimated for these three time intervals.

OTHER OUTCOMES:
Glucose control at start of the study | At Baseline
  In all participants, Hemoglobin A1c (HbA1c) is measured before the start of the study and comparisons are made between the three treatment groups regarding mean HbA1c and how dispersed the data is in relation to the mean (standard deviation). A lower HbA1c means a better glucose control and a lower standard deviation means less variability within the group.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Adolfsson, MD PhD, Principal Investigator — Västra Götalandsregionen, Gothenburg University
Locations (1):
- The hospital of Halland Kungsbacka, Kungsbacka, Region of Halland, Sweden

IPD SHARING:
Plan to Share IPD: No